CLINICAL TRIAL: NCT02472717
Title: Clinical Evaluation of Psoriatic Arthritis Treated With Liraglutide. The PLAQUE Study: Psoriatic Arthritis Treated With Liraglutide Therapy: a QUality of Life and Efficacy Study
Brief Title: Psoriatic Arthritis Treated With Liraglutide Therapy: a QUality of Life and Efficacy Study
Acronym: PLAQUE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1150-8501
Record Dates: First submitted 2015-05-27; First posted 2015-06-16 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2015-06

CONDITIONS: Psoriatic Arthritis; Psoriasis; Impaired Glucose Tolerance; Type 2 Diabetes
Keywords: liraglutide, GLP-1 receptor agonists
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional arm (Experimental): liraglutide 0.6mg sc daily for 1 week, 1.2mg sc daily for 11 weeks
  Interventions: Drug: liraglutide
- Placebo arm (Placebo Comparator): Placebo sc daily for 12 weeks, volume titration at week 2 to mirror liraglutide arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: liraglutide — Liraglutide 0.6mg sc daily for 1 week, 1.2mg sc daily for 11 weeks
  Other Names: Victoza
  Arms: Interventional arm
Other: Placebo — Placebo sc daily for 12 weeks, volume titration at week 2 to mirror liraglutide arm
  Arms: Placebo arm

SUMMARY:
Exploratory, double-blind randomized, placebo-controlled, Phase II study to evaluate the effect(s) of short-term administration of liraglutide, a GLP-1R (glucagon-like peptide-1 receptor) agonist on joint and skin inflammation in patients with active Psoriatic Arthritis.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether short-term (12-week) administration of the GLP-1R agonist, liraglutide, will improve joint and skin swelling in patients with active Psoriatic Arthritis compared to placebo.

Background: Psoriatic Arthritis is a systemic inflammatory T-cell disorder affecting the joints and spine, and is associated with an elevated risk for Type 2 Diabetes and Cardiovascular Disease. In addition to classical effects on glycemic-lowering, GLP-1R agonists are anti-diabetes agents which also have anti-inflammatory properties that may be clinically useful for patients with inflammatory diseases, particularly those with co-morbid metabolic disease. While a few small exploratory studies in patients with psoriasis have demonstrated that GLP-1R agonists reduce the severity of skin plaques, dedicated prospective, randomized mechanistic studies evaluating potential mechanisms by which GLP-1R agonists exert anti-inflammatory action(s) in humans with inflammatory disease is lacking.

Objectives: Primary objective is to evaluate the clinical efficacy of short-term liraglutide (GLP-1R agonist) administration on the severity of joint and skin inflammation in patients with active Psoriatic Arthritis. Secondary objectives are to determine whether short-term liraglutide administration in patients with active psoriatic arthritis will 1) modify the degree of impaired glucose tolerance, underlying b-cell function and cardiovascular risk factor profiles, 2) improve patient-centered outcomes such as quality of life and functionality, 3) modify specific sub-populations of T-cells and affect their differentiation and activation, and 4) modify activation of circulating immune cells, pro-inflammatory cytokines, and hormones.

Design: Double-blind, randomized, placebo-controlled trial, Phase II.

Patient population: 34 patients between with active Psoriatic Arthritis meeting CASPAR (ClASsification criteria for Psoriatic ARthritis).

Intervention: Participants will be randomized (1:1) to liraglutide (1.2 mg sc daily) or to placebo (sc daily) for 12 weeks.

Endpoints: The primary endpoint of this study will be the proportion of patients who experience a 20% ACR (American College of Rheumatology) improvement response following liraglutide therapy as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active psoriatic arthritis (3 tender and swollen joints) meeting CASPAR study group criteria

Exclusion Criteria:

* BMI > 35 kg/m2
* Uncontrolled diabetes, HbA1c > 10.5%
* Current biological treatment for any inflammatory disorder within the past three months
* renal dysfunction (eGFR < 50 ml/min/1.73m or macroalbuminuria >300mg)
* hepatic dysfunction (AST (aspartate aminotransferase), ALT (alanine aminotransferase), Total bilirubin > 3 times upper limit of normal)
* history of pancreatitis or personal or family history of medullary thyroid cancer, c-cell hyperplasia, or MEN-2 syndrome
* current pregnancy or current breast feeding
* use of DPP-4 (dipeptidyl peptidase-4 inhibitor) or GLP-1 receptor agonist within 2 months (washout is permitted)
* drug or alcohol dependence
* resting tachycardia > 100 bpm or conduction abnormalities associated with tachycardia
* current enrollment in any other clinical trial
* symptomatic gastroparesis
* concomitant serious medical conditions
* all medication for the treatment of Psoriatic Arthritis such as MTX (methotrexate) < 25 mg, LFN (leflunomide) < 20 mg, and NSAIDs (non-steroidal anti-inflammatory drugs) will have been used at stable doses for at least 4 weeks, having been initiated at least 3 months prior to study start (8 weeks before screening, 4 weeks before baseline) for MTX and LFN and at least 4 weeks for NSAIDs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The change in the proportion of patients achieving an ACR 20% improvement response in patients with psoriatic arthritis receiving liraglutide for 12 weeks compared to placebo | Baseline to 12 weeks, liraglutide compared to placebo
  Proportion of patients achieving an ACR (American College of Rheumatology) 20% improvement response. ACR 20 is a composite rheumatological endpoint which includes swollen joint count, tender joint count, pain, physician global assessment, patient global assessment, HAQ (health assessment questionnaire), CRP (c reactive protein).

SECONDARY OUTCOMES:
The change in the psoriasis area and severity index (PASI) in patients with psoriatic arthritis receiving liraglutide for 12 weeks compared to those receiving placebo | Baseline to 12 weeks
The change in quality of life measured by validated quality of life questionnaires in patients with psoriatic arthritis receiving liraglutide for 12 weeks compared to those receiving placebo | Baseline to 12 weeks
The change in glucose tolerance in patients with psoriatic arthritis with glucose intolerance at baseline who receive liraglutide for 12 weeks compared to those receiving placebo | Baseline to 12 weeks
The effect(s) of liraglutide on cardiovascular disease risk factors in patients with psoriatic arthritis receiving liraglutide for 12 weeks compared to those receiving placebo | Baseline to 12 weeks
  Cardiovascular disease risk factors (Systolic blood pressure, cholesterol profiles, CRP, body weight, waist circumference)
The effect(s) of liraglutide on the enumeration of circulating T-cell subpopulations, and on activation of circulating T-cell subpopulations | Baseline to 12 weeks
  Multi-parameter phospho flow cytometry analysis of T-cell differentiation and activation of peripheral blood

OTHER OUTCOMES:
The effect of liraglutide on levels of infiltrating dermal T cells and cytokines in psoriatic skin plaques from patients with psoriatic arthritis receiving liraglutide therapy for 12 weeks compared to those receiving placebo | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, The Centre for Prognosis Studies in the Rheumatic Diseases (CPSRD), University of Toronto, Toronto, Ontario, Canada